CLINICAL TRIAL: NCT03924687
Title: A Randomized Controlled Trial Evaluating the Effectiveness of an Acceptance and Commitment Therapy-Based Bibliotherapy Intervention Among Adults Living With Chronic Pain
Brief Title: Evaluating the Effectiveness of an ACT-Based Bibliotherapy Intervention Among Adults Living With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Dr. Frédérick Dionne, Ph.D., Associate Professor, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER-15-215-07.23
Record Dates: First submitted 2019-04-08; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Chronic Pain
Keywords: chronic pain; Acceptance or Commitment Therapy (ACT); self-help; pain-related disability; psychological inflexibility; depression; pain acceptance; bibliotherapy
MeSH Terms: conditions — Chronic Pain; Depression | interventions — Bibliotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT group (Experimental): ACT group: participants receiving the 8-week bibliotherapy intervention based on Acceptance and Commitment Therapy
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT) bibliotherapy for chronic pain
- control group (No Intervention): Wait-list control condition: participants placed on a wait-list (and receiving the intervention following the 9 week duration of the intervention)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) bibliotherapy for chronic pain — The intervention consisted of the book "Libérez-vous de la douleur par la méditation et l'ACT" (Dionne, 2014) and a participant workbook, along with two phone calls of approximately 15 minutes each and weekly e-mails presenting the week's content. Participants also had access to audio meditation exercises on the book's website (http://liberezvousdeladouleur.com/meditations/).
  Arms: ACT group

SUMMARY:
Chronic pain has a significant impact on the physical and psychological functioning of those living with this condition. It is now recognized that Acceptance and Commitment Therapy (ACT) is an effective intervention in managing chronic pain; however, several barriers limit its accessibility.

The current study aims to evaluate the effectiveness of an eight-week bibliotherapy-type self-administered psychological intervention with minimal therapeutic contact, based on ACT, in the management of chronic pain.

This study is a randomized controlled trial with two groups (one experimental group and one wait-list control group). Participants will be randomly assigned to each condition and measures will be taken at pretest, posttest and three months following the intervention.

DETAILED DESCRIPTION:
The purpose of this randomized controlled trial was to assess the effectiveness of an eight-week self-administered intervention program (bibliotherapy) based on Acceptance and Commitment Therapy with minimal therapeutic support in the management of chronic pain.

This study was based on the following hypotheses. In comparison to the control group, from pre to post, the self-help program will:

1. significantly reduce pain-related disability (primary variable);
2. improve depressive symptoms related to CP (secondary variable);
3. increase the level of pain acceptance;
4. reduce psychological inflexibility linked to painful symptoms (process variables).

   It was also expected that:
5. the improvements would be maintained at three-month follow-up;
6. participants would have an overall impression of a positive change following the intervention.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years of age or older
* having suffered from daily pain for more than three months
* having reading and writing abilities in French equivalent or superior to grade 8
* having access to Internet at home and having a valid e-mail address
* not having previously completed an ACT-type psychotherapy, not having practiced mindfulness meditation regularly and not having read a bibliotherapy on ACT for pain
* having stable medication for at least one month, if applicable.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-03-28 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Pain-related disability | Change from week 1 to week 9
  Brief Pain Inventory (BPI; Interference subscale; Cleeland & Ryan 1994; Poundja, Fikretoglu, Guay, & Brunet 2007; Tyler, Jensen, Engel, & Schwartz 2002)
Change in Pain-related disability | Change from week 9 and week 21 (ACT group only)
  Brief Pain Inventory (BPI; Interference subscale; Cleeland & Ryan 1994; Poundja, Fikretoglu, Guay, & Brunet 2007; Tyler, Jensen, Engel, & Schwartz 2002)

SECONDARY OUTCOMES:
Change in Depressive symptoms | Change from week 1 to week 9
  The Beck Depression Inventory (BDI - Short Form: Beck, Rial, & Rickels 1974)
Change in Depressive symptoms | Change from week 9 and week 21 (ACT group only)
  The Beck Depression Inventory (BDI - Short Form: Beck, Rial, & Rickels 1974)
Change in Pain acceptance | Change from week 1 to week 9
  Chronic Pain Acceptance Questionnaire (CPAQ-8: Fish, McGuire, Hogan, Morrison, & Stewart 2010). The CPAQ-8 is an 8-item measure that evaluates acceptance of pain according to two sub-scales: activity engagement and pain willingness. Items are rated on a Likert scale from 0 = never true to 6 = always true. Total scores range from 0 to 48 and higher scores reflect greater acceptance of pain.
Change in Pain acceptance | Change from week 9 and week 21 (ACT group only)
  Chronic Pain Acceptance Questionnaire (CPAQ-8: Fish, McGuire, Hogan, Morrison, & Stewart 2010). The CPAQ-8 is an 8-item measure that evaluates acceptance of pain according to two sub-scales: activity engagement and pain willingness. Items are rated on a Likert scale from 0 = never true to 6 = always true. Total scores range from 0 to 48 and higher scores reflect greater acceptance of pain.
Change in Psychological inflexibility | Change from week 1 to week 9
  Psychological Inflexibility in Pain Scale (PIPS; Wicksell, Lekander, et al. 2010). The PIPS is composed of 12 items that evaluate two dimensions: avoidance and cognitive fusion. Items are rated on a Likert scale from 1 = never true to 7 = always true, to evaluate the level of inflexibility associated to pain. Scores range from 12 to 84, with higher scores revealing greater psychological inflexibility.
Change in Psychological inflexibility | Change from week 9 and week 21 (ACT group only)
  Psychological Inflexibility in Pain Scale (PIPS; Wicksell, Lekander, et al. 2010). The PIPS is composed of 12 items that evaluate two dimensions: avoidance and cognitive fusion. Items are rated on a Likert scale from 1 = never true to 7 = always true, to evaluate the level of inflexibility associated to pain. Scores range from 12 to 84, with higher scores revealing greater psychological inflexibility.
Participants' impression of change | week 21
  Patient Global Impression of Change (PGIC: Guy et al. 1976)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hann, K. E. J., & McCracken, L. M. (2014). A systematic review of randomized controlled trials of Acceptance and Commitment Therapy for adults with chronic pain: Outcome domains, design quality, and efficacy. Journal of Contextual Behavioral Science, 3(4), 217-227. http://dx.doi.org/http://dx.doi.org/10.1016/j.jcbs.2014.10.001
- [Background] Hughes LS, Clark J, Colclough JA, Dale E, McMillan D. Acceptance and Commitment Therapy (ACT) for Chronic Pain: A Systematic Review and Meta-Analyses. Clin J Pain. 2017 Jun;33(6):552-568. doi: 10.1097/AJP.0000000000000425. PMID 27479642
- [Background] Boulanger, A., Charbonneau, C., Choinière, M., Laliberté, J., & St-Hilaire, F. (2015). Renforcer les services de première ligne, développer les connaissances et les compétences des patients et des professionnels de la santé afin de mieux prévenir et traiter la douleur chronique.
- [Background] Hogg MN, Gibson S, Helou A, DeGabriele J, Farrell MJ. Waiting in pain: a systematic investigation into the provision of persistent pain services in Australia. Med J Aust. 2012 Apr 2;196(6):386-90. doi: 10.5694/mja12.10140. PMID 22471539
- [Background] Jamison RN, Gintner L, Rogers JF, Fairchild DG. Disease management for chronic pain: barriers of program implementation with primary care physicians. Pain Med. 2002 Jun;3(2):92-101. doi: 10.1046/j.1526-4637.2002.02022.x. PMID 15102155
- [Background] Hayes, S. C., Strosahl, K. D., & Wilson, K., G. (2012). Acceptance and commitment therapy : the process and practice of mindful change (2nd ed.). New York: Guilford Press.
- [Derived] Veillette J, Martel ME, Dionne F. A randomized controlled trial evaluating the effectiveness of an acceptance and commitment therapy-based bibliotherapy intervention among adults living with chronic pain. Can J Pain. 2019 Nov 26;3(1):209-225. doi: 10.1080/24740527.2019.1678113. eCollection 2019. PMID 35005411